CLINICAL TRIAL: NCT03496883
Title: Recombinant Factor VIIa (rFVIIa) for Acute Hemorrhagic Stroke Administered at Earliest Time (FASTEST) Trial
Brief Title: Recombinant Factor VIIa (rFVIIa) for Hemorrhagic Stroke Trial
Acronym: FASTEST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Joseph Broderick, MD (Other)
Collaborators: Novo Nordisk A/S (Industry); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Joseph Broderick, MD, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCincinnatifastest; 1U01NS110772-01 (NIH); 2019-003722-25 (EudraCT Number); U1111-1201-0087 (Other: Universal Trial Number)
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded study medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recombinant Activated Factor VII (rFVIIa) (Active Comparator): rFVIIa given as IV injection over 2 minutes within 120 minutes of stroke onset
  Interventions: Biological: Recombinant Activated Factor VII (rFVIIa)
- Placebo (Placebo Comparator): Matching placebo given as IV injection over 2 minutes within 120 minutes of stroke onset
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Recombinant Activated Factor VII (rFVIIa) — Participants will be randomized in a double-blinded fashion to rFVIIa 80 µg/kg dose (maximum 10 mg dose) or matching placebo. Participants in both arms will receive best standard therapy as per published AHA Guidelines for ICH, including a target systolic blood pressure of 140 mm Hg.
  Other Names: NovoSeven; NiaStase
  Arms: Recombinant Activated Factor VII (rFVIIa)
Biological: Placebo — Participants will be randomized in a double-blinded fashion to rFVIIa 80 µg/kg dose (maximum 10 mg dose) or matching placebo. Participants in both arms will receive best standard therapy as per published AHA Guidelines for ICH, including a target systolic blood pressure of 140 mm Hg.
  Arms: Placebo

SUMMARY:
The objective of the rFVIIa for Acute Hemorrhagic Stroke Administered at Earliest Time (FASTEST) Trial is to establish the first treatment for acute spontaneous intracerebral hemorrhage (ICH) within a time window and subgroup of patients that is most likely to benefit. The central hypothesis is that rFVIIa, administered within 120 minutes from stroke onset with an identified subgroup of patients most likely to benefit, will improve outcomes at 180 days as measured by the Modified Rankin Score (mRS) and decrease ongoing bleeding as compared to standard therapy.

DETAILED DESCRIPTION:
The investigators will perform a global, Phase III, randomized, double-blind controlled trial of rFVIIa plus best standard therapy vs. placebo and best standard therapy alone. The investigators will include participants with a volume of ICH ≥ 2 and < 60 cc, no more than a small volume of intraventricular hemorrhage (IVH) (IVH score ≤ 7), age ≥ 18 and ≤ 80, Glasgow Coma Scale of ≥ 8, and treated within 120 minutes from stroke onset. To minimize time-to-treatment, the study will use emergency research informed consent procedures (including exception from informed consent (EFIC) in the United States) and mobile stroke units (MSUs), with a goal of ½ of participants treated within 90 minutes, as accomplished in the NINDS t-PA trials. The FASTEST Trial will include approximately 100 hospital sites and at least 15 MSUs in the NINDS-funded StrokeNet and key global institutions with large volumes of ICH patients and the ability to treat them within 120 minutes of stroke onset. Recruitment of 860 participants over 3½ years is planned. Countries participating in the trial include the United States, Canada, Japan, Germany, Spain, and the United Kingdom. Involving other countries may be possible in the future depending upon recruitment needs.

Participants will be randomized in a double-blinded fashion to rFVIIa 80 µg/kg dose (maximum 10 mg dose) or placebo. Participants in both arms will receive best standard therapy as per published AHA Guidelines for ICH, including a target systolic blood pressure of 140 mm Hg. The primary outcome (ordinal mRS with the following categories: 0-2, 3, and 4-6) will be determined at 180 days, but participants will be followed by remote assessment at 30 days and 90 days. To measure growth of ICH, all participants will have a standard of care baseline non-contrast CT of the head and a repeat scan at 24 hours. Centralized volumetric measurements of ICH, IVH, and edema will be performed for both time points.

Novo Nordisk A/S will manufacture and supply rFVIIa as a research medication for use in the FASTEST Trial. Novo Nordisk A/S will also manufacture and supply matching placebo that is identical to rFVIIa in appearance and administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years, inclusive
2. Patients with spontaneous ICH
3. Able to treat with study medication (rFVIIa/placebo) within 120 minutes of stroke onset or last known well
4. Efforts to obtain informed consent per EFIC guidelines (U.S.) or adherence to country-specific emergency research informed consent regulations (Canada, Germany, Spain, U.K., Japan)

Exclusion Criteria:

1. Score of 3 to 7 on the Glasgow Coma Scale
2. Secondary ICH related to known causes (e.g., trauma, aneurysm, arteriovenous malformation (AVM), oral anticoagulant use (vitamin K antagonists or novel oral anticoagulants) within the past 7 days, coagulopathy, etc.)
3. ICH volume < 2 cc or ≥ 60 cc
4. Blood filling 2/3 or more of one lateral ventricle of the brain, OR, blood filling at least 1/3 of both lateral ventricles.
5. Pre-existing disability (mRS > 2)
6. Symptomatic thrombotic or vaso-occlusive disease in past 90 days (e.g., cerebral infarction, myocardial infarction, pulmonary embolus, deep vein thrombosis, or unstable angina)
7. Clinical or EKG evidence of ST elevation consistent with acute myocardial ischemia
8. Brainstem location of hemorrhage (patients with cerebellar hemorrhage may be enrolled)
9. Refusal to participate in study by patient, legal representative, or family member
10. Known or suspected thrombocytopenia (unless current platelet count documented above 50,000/μL)
11. Unfractionated heparin use with abnormal PTT
12. Pro-coagulant drugs within 24 hours prior to patient enrollment into the FASTEST trial (example, tranexamic acid or aminocaproic acid)
13. Low-molecular weight heparin use within the previous 24 hours
14. Recent (within 90 days) carotid endarterectomy or coronary or cerebrovascular angioplasty or stenting
15. Advanced or terminal illness or any other condition the investigator feels would pose a significant hazard to the patient if rFVIIa were administered
16. Recent (within 30 days) participation in any investigational drug or device trial or earlier participation in any investigational drug or device trial for which the duration of effect is expected to persist until to the time of FASTEST enrollment
17. Planned withdrawal of care or comfort care measures
18. Patient known or suspected of not being able to comply with trial protocol (e.g., due to alcoholism, drug dependency, or psychological disorder)
19. Known or suspected allergy to trial medication(s), excipients, or related products
20. Contraindications to study medication
21. Previous participation in this trial (previously randomized)
22. Females of childbearing potential who are known to be pregnant or within 12 weeks post-partum and/or lactating at time of enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 180 days
  Ordinal distribution with the following steps: 0-2, 3, 4-6

SECONDARY OUTCOMES:
mRS | 180 days
  Utility-weighted
mRS | 180 days
  Score of 0-2
EQ-5D | 180 days
  Quality of life scale
Change in the volume of ICH and ICH+IVH | Between baseline CT and 24-hour CT
  As measured by non-contrast CT of the head
mRS | 90 days
  Ordinal distribution
EQ-5D | 90 days
  Quality of life scale
mRS | 180 days
  Ordinal distribution

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Broderick, MD, Principal Investigator — University of Cincinnati
Locations (88):
- United States (51):
  - University of Alabama Hospital, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Kaiser Permanente Baldwin Park Medical Center, Baldwin Park, California
  - Mills Peninsula Medical Center, Burlingame, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Kaiser Permanente South Bay Medical Center, Harbor City, California
  - UCSD Health La Jolla, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC Irvine Medical Center,, Orange, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - UC Davis Medical Center, Sacramento, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - UF Health Shands Hospital, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - M Health Fairview Ridges Hospital,, Burnsville, Minnesota
  - M Health Fairview Southdale Hospital, Edina, Minnesota
  - M Health Fairview St. John's Hospital, Maplewood, Minnesota
  - M Health Fairview University of Minnesota Medical Center Hospital,, Minneapolis, Minnesota
  - Mayo Clinic Saint Marys Campus, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai West, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina University Hospital, Charleston, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - VCU Medical Center, Richmond, Virginia
- Canada (8):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - University of Montreal Hospital, Montreal, Quebec
- Germany (5):
  - University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg
  - Clinic Frankfurt Hoechst, Frankfurt am Main, Hesse
  - University Hospital Augsburg, Augsburg
  - Charite University Medicine Berlin, Berlin
  - University Hospital Tuebingen, Tübingen
- Japan (14):
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Kyushu Medical Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Kagoshima City Hospital, Kagoshima
  - Kobe City Medical Center General Hospital, Kobe
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Iwate Prefectural Central Hospital, Morioka
  - Niigata City General Hospital, Niigata
  - KMU University Hospital, Osaka
  - NHO Osaka National Hospital, Osaka
  - Nakamura Memorial Hospital, Sapporo
  - Jichi Medical University Hospital, Shimotsuke
  - Kyorin University Hospital, Tokyo
  - Toranomon Hospital, Tokyo
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Vall d'Hebron University Hospital (VHUH), Horta, Barcelona
  - Bellvitge University Hospital,, L'Hospitalet de Llobregat, Barcelona
  - Santa Creu and Sant Pau Hospital, Barcelona, Catalonia
  - Girona University Hospital, Girona, Catalonia
  - Arnau de Vilanova University Hospital, Lleida, Catalonia
- United Kingdom (4):
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Results to be reported on ClinicalTrials.gov, and trial database prepared for NINDS for sharing with other investigators
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available 12 months after publication of primary results
Access Criteria: Approval by NINDS

REFERENCES:
- [Derived] Broderick JP, Naidech AM, Elm JJ, Toyoda K, Dowlatshahi D, Demchuk AM, Khatri P, Steiner T, Bath PM, Audebert HJ, Vagal A, Yoshimura S, Mayer SA, Wang LL, Sabagha N, Mocco JD, Molina C, Aviv R, Stinson E, Quadri SA, Carrozzella J, Huynh T, Phan A, Beall J, Davis I, Sakai N, Ohta T, Yokosawa M, Hara T, Sangha N, Morita K, Dominc Tse MY, Streib CD, Miyashita F, Silva Y, Nagakane Y, Gheorghiu T, Sun CH, Hirano T, Poli S, Izumo T, Fukuda-Doi M, Ihara M, Koga M, Buck B, Walsh KB, Spokovny I, Grotta JC; FASTEST Investigators. Recombinant factor VIIa versus placebo for spontaneous intracerebral haemorrhage within 2 h of symptom onset (FASTEST): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet. 2026 Feb 4:S0140-6736(26)00097-8. doi: 10.1016/S0140-6736(26)00097-8. Online ahead of print. PMID 41653933
- [Derived] Yu W, Alexander MJ. Spontaneous intracerebral hemorrhage: Recent advances and critical thinking on future clinical trial design. Chin Med J (Engl). 2024 Dec 20;137(24):2899-2906. doi: 10.1097/CM9.0000000000003408. Epub 2024 Dec 10. No abstract available. PMID 39654449
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Naidech AM, Grotta J, Elm J, Janis S, Dowlatshahi D, Toyoda K, Steiner T, Mayer SA, Khanolkar P, Denlinger J, Audebert HJ, Molina C, Khatri P, Sprigg N, Vagal A, Broderick JP. Recombinant factor VIIa for hemorrhagic stroke treatment at earliest possible time (FASTEST): Protocol for a phase III, double-blind, randomized, placebo-controlled trial. Int J Stroke. 2022 Aug;17(7):806-809. doi: 10.1177/17474930211042700. Epub 2021 Sep 5. PMID 34427473
- See also: Related Info — https://www.nihstrokenet.org/trials/fastest/home